CLINICAL TRIAL: NCT05938556
Title: The Impact of a Multicenter Randomized Control Trial of Hybrid Synchronous-Asynchronous Virtual Group Coaching on Burnout and Retention in Advanced Practice Providers
Brief Title: Coaching for Advanced Practice Providers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Children's Healthcare of Atlanta (Other); University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Zahidee (Saidie) Rodriguez, Assistant Professor, Emory University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00005675
Record Dates: First submitted 2023-06-08; First posted 2023-07-10 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Burnout, Professional
Keywords: Advanced Practice Providers; APPs; Coaching; Healthcare provider; Nurse burnout; Wellness
MeSH Terms: conditions — Burnout, Professional | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to receive either four months of group coaching or treatment as usual. After fourth months of the assigned treatment, the two arms will switch for another four months of either group coaching or treatment as usual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Coaching Program (Experimental): The study intervention is a hybrid asynchronous-synchronous group coaching treatment that will occur over four months. Participants will be given access to a members-only, web-based platform to access the intervention.
  Interventions: Behavioral: hybrid asynchronous-synchronous group coaching program
- Usual Treatment (Placebo Comparator): This group will participate in the study intervention following a 4-month waitlist/control group.
  Interventions: Other: treatment as usual group (TAU)

INTERVENTIONS:
Behavioral: hybrid asynchronous-synchronous group coaching program — A hybrid asynchronous-synchronous program. The synchronous part has two weekly recorded live group coaching calls for four months. The asynchronous consist of 1) on-demand replies to recorded coaching calls, 2) Self-coaching through weekly self-study modules and worksheets, and 3) written Ask A Coach. Content modified per needs of APPs by a physician, a certified coach, and an APP who is also a Co-I. The curriculum has weekly themes that build. Month-1 consists of 1) Introduction to the Model, 2) How to Feel Better, 3) Defining Your Purpose, and 4) Living Your Purpose. Month-2 consists of 1) Growth Mindset, 2) Welcoming Feedback and Assessment Bias, 3) Feeling Valued and Belonging, and 4) How to Deal with Hidden Expectations. Month-3 consists of 1) Imposter Syndrome, 2) Perfectionism, 3) Approval Addiction, and 4) How to Change Your Thoughts. Month-4 consists of 1) How to deal with Ambiguity, 2) Confidence, 3) Self-Appreciation and Self-Compassion, and 4) Celebrate the New You.
  Other Names: group coaching program
  Arms: Group Coaching Program
Other: treatment as usual group (TAU) — The treatment as usual group will consist of any structural or programmatic interventions, resources, lectures, curriculum, etc. offered at the participants' hospital of employment. Thus, this active control is designed to represent a best-case alternative to group coaching, making it a more rigorous form of control. Participants randomly assigned to TAU will also continue any structural or programmatic interventions or resources they were previously participating in.
  Other Names: TAU
  Arms: Usual Treatment

SUMMARY:
This study aims to determine if online coaching is feasible in advanced practice providers (APP) and can impact burnout.

The study will recruit APPs from Children's Healthcare of Atlanta (CHOA), Emory, Colorado University (CU), and their affiliate hospitals through online consent sent via email. Interventions will include online video coaching, written coaching, and self-coaching through self-study material.

DETAILED DESCRIPTION:
The purpose of this study is to determine the feasibility of establishing a coaching program directed toward Advanced Practice Providers (APPs), to determine the generalizability of tools shown to relieve physician burnout in the population of APPs, and to advance research in the field of healthcare wellness.

The coaching group will have a curriculum of self-study modules, pre-recorded webinars, and worksheets. The coaching group will also have access to two live group calls per week as well as an online forum to receive anonymously written coaching. After four months, participants will be switched to the other group, so that each participant is exposed to treatment but at separate times. At the completion of each intervention time point, participants will fill out a post-study survey.

ELIGIBILITY:
Inclusion Criteria:

* Advanced Practice Providers (nurse practitioners, physician assistants, certified midwife nurses, certified registered nurse anesthetists, anesthesiology assistants, and clinical nurse specialists) at Children's Healthcare of Atlanta, Emory University, and CU and its affiliate hospitals.
* Pregnant women will be included in this population, though this inclusion is incidental.

Exclusion Criteria:

* adults unable to consent,
* individuals who are not adults,
* prisoners,
* cognitively impaired or individuals with impaired decision-making capacity and
* individuals who do not clearly understand English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2023-07-14 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Burnout | Baseline, 4 months, 9 months
  Burnout as defined by the Maslach Burnout Inventory (MBI). The Maslach burnout inventory (MBI) is a 22-item measurement of worker burnout that assesses emotional exhaustion (EE), depersonalization (DP), and personal fulfillment (PF) domains. Possible scores range from 0-6 on a Likert scale for each item. Scores of EE ≥ 27 points, DP ≥ 10, and PF <33 would indicate a high degree of burnout. Scores of EE≤18 points, DP≤5 points, and PF≥40 points would indicate a low degree of burnout.
Change in the percentage of participants that accept the program course | Baseline, 4 months, 9 months
  Data collection will be at baseline, month 4, and month 9 for both groups.
Percentage of participants who watch program calls | 4 month or 9 months
  Number of participants who watch program calls. Data collection will only be at the end of participation Group Coaching Program.
Change in the percentage of participants that complete >50% of self-study worksheets | 4 month or 9 months
  Number of participants who complete >50% of self-study worksheets. Data collection will only be at the end of participation Group Coaching Program.
Change in the percentage of participants that use the Ask A Coach Forum at least once | 4 month or 9 months
  Percentage of participants that use the Ask A Coach Forum at least once. Data collection will only be at the end of participation Group Coaching Program.
Change in the rate of participation in the program | Baseline, 4 months, 9 months
  Percentage of participants that complete the outcome measures (pre/post surveys). Data collection will be at month 4 and month 9 for both groups.

SECONDARY OUTCOMES:
Change in Trauma Symptoms of Discrimination Scale | Baseline, 4 months, 9 months
  This two-part scale measures the experiences of discrimination using trauma symptoms. Part 1 includes 21 questions where the participant can respond to agree or disagree with the statement using Likert scale response options. Part 2 of the scale allows the respondent to allocate what percentage of their identity they experience discrimination on (i.e. race/ethnicity: 70%, disability: 20 %, and gender: 10%).
Change in Self-Compassion | Baseline, 4 months, 9 months
  Self-Compassion as defined by Neff's Self Compassion Score Short Form is a 12-item measurement of self-compassion. Possible scores range from 0-6 on a Likert scale for each item, where the higher scale scores indicate greater self-compassion. Scores of 1.0- 2.49 are considered to be low, between 2.5-3.5 to be moderate, and 3.51-5.0 to be high.
Change in Moral Injury | Baseline, 4 months, 9 months
  Moral Injury as defined by the Moral Injury Symptom Scale for Health Professions. (MISS-HP) is a 10-item measurement of moral injury. Possible scores range from 0-5 on a Likert scale for each item, where the higher scale scores indicate greater moral injury. Scores >35 (on a possible score range of 10 to 100) are considered high for moral injury symptoms causing moderate to extreme problems with family, social, and occupational functioning.
Change in the Young's Imposter Syndrome Symptoms Scale | Baseline, 4 months, 9 months
  Imposter Syndrome as defined by Young's Imposter Syndrome Symptoms Scale. (YISS) is an 8-item measurement of imposter syndrome. Scoring is yes/no where a score of >5/8 is felt to be positive for imposter syndrome.
Change in the intention to leave | Baseline, 4 months, 9 months
  Intent-to-leave is defined by a single-item question, on a 3-point Likert scale, where the higher the score reflects more intention to leave the current position. Followed by a single multiple-choice question as to why the participant is leaving.
Change in Loneliness | Baseline, 4 months, 9 months
  Loneliness as defined by the University of California, Los Angeles (UCLA) 3-item Loneliness Scale. It is a 3-item measure of relational connectedness, social connectedness, and self-perceived isolation. Items are measured on a 3-point scale where a score range of 3-5 is "not lonely" and a score range of 6-9 is "lonely".
Change in Self Reflection and Insight Scale | Baseline, 4 months, 9 months
  Self-reflection and insight as defined by Self Reflection and Insight Short Scale (SIRSS). It is a 12-point item measurement of the capacity to reflect on oneself and to think about one's thoughts, experiences, and actions on a 7-point Likert scale, where higher scores reflect more inspection, evaluation and perception of thoughts, beliefs, feelings, and behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Zahidee (Saidie) Rodriguez, MD, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - University of Colorado, Denver, Colorado
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Emory Healthcare System, Atlanta, Georgia
  - Emory University, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
Investigators will share all of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Proposals should be directed to rodriguezz@kidsheart.com with a signed data access agreement, for up to 5 yrs (example 2 language)